CLINICAL TRIAL: NCT01286987
Title: A Phase 1, First In Human, Single-arm, Open-label Study Of Once A Day, Orally Administered Talazoparib (Bmn 673) In Patients With Advanced Or Recurrent Solid Tumors
Brief Title: Study of Talazoparib, a PARP Inhibitor, in Patients With Advanced or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PRP-001; 2010-023062-40 (EudraCT Number); C3441007 (Other: Alias Study Number)
Record Dates: First submitted 2011-01-26; First posted 2011-02-01 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-06

CONDITIONS: Advanced or Recurrent Solid Tumors; Breast Neoplasms; Ovarian Cancer, Epithelial; Ewing Sarcoma; Small Cell Lung Carcinoma; Prostate Cancer; Pancreas Cancer
Keywords: BRCA1 Protein; BRCA2 Protein
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ovarian Epithelial; Sarcoma, Ewing; Small Cell Lung Carcinoma; Prostatic Neoplasms; Pancreatic Neoplasms; Fanconi Anemia, Complementation Group D1 | interventions — talazoparib

ARMS (1):
- Talazoparib (Experimental)
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Oral capsule with multiple dosage forms given once daily
  Other Names: BMN 673; MDV3800

SUMMARY:
This is a single-arm, open-label study to assess the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of talazoparib in patients with advanced tumors with DNA-repair pathway deficiencies. There will be 2 parts to the study: a dose escalation phase in which the maximum tolerated dose will be defined, and a dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, unresectable, locally advanced or metastatic solid tumor
* Must have available archived tumor tissue (formalin-fixed paraffin-embedded) [FFPE].
* 18 years of age or older.
* Have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST, v1.1) or increased CA-125 (ovarian cancer) or PSA (prostate cancer) and/or CA 19-9 (pancreatic cancer).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Have adequate organ function
* Able to take oral medications.
* Willing and able to provide informed consent.
* Sexually active patients must be willing to use an acceptable method of contraception.
* Females of childbearing potential must have a negative serum pregnancy test at screening.
* Willing and able to comply with all study procedures.

Part 2 Dose Expansion Tumor Types:

* Breast and ovarian cancer patients with deleterious or pathogenic BRCA mutations who have received no more than 4 prior regimens for metastatic disease.
* Prostate or pancreatic cancer patients with deleterious or pathogenic BRCA mutations who have received no more than 2 prior regimens for metastatic disease.
* Small cell lung cancer (SCLC) patients who have received no more than one prior regimen for SCLC.
* Ewing's sarcoma patients who have received no more than 3 prior regimens for metastatic disease.

Exclusion Criteria:

* Part 2 Expansion: Prior treatment with a PARP inhibitor.
* Has history of central nervous system (CNS) metastasis.

  * Exception: In patients with SCLC, history of adequately treated brain metastasis who do not require corticosteroids for management of CNS symptoms.
* Has had major surgery within 28 days before Cycle 1, Day 1.
* Has active peptic ulcer disease.
* Active gastrointestinal tract disease with malabsorption syndrome.
* Pregnant or breastfeeding at screening or planning to become pregnant (in each case, either oneself or one's partner) at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-01-03 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2017-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Medical Director, Study Director — Medivation, Inc.
Locations (15):
- United States (14):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Virginia G. Piper Cancer Center Research Pharmacy, Scottsdale, Arizona
  - (IRB# 12-000131) Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Westwood Bowyer Clinic, Peter Morton Medical Building, Los Angeles, California
  - Santa Monica - UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - IU Health Bloomington Hospital, Bloomington, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted in two parts: Part 1 was dose escalation phase (to determine the maximum tolerated dose [MTD]) and Part 2 was the dose expansion phase conducted at MTD determined in Part 1. Participants were different in both of the Parts.
Groups:
- Part 1: Talazoparib 25 mcg/Day: Participants received talazoparib capsules at a dose of 25 microgram per day (mcg/day) once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 50 mcg/Day: Participants received talazoparib capsules at a dose of 50 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 100 mcg/Day: Participants received talazoparib capsules at a dose of 100 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 200 mcg/Day: Participants received talazoparib capsules at a dose of 200 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 400 mcg/Day: Participants received talazoparib capsules at a dose of 400 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 600 mcg/Day: Participants received talazoparib capsules at a dose of 600 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 900 mcg/Day: Participants received talazoparib capsules at a dose of 900 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 1000 mcg/Day: Participants received talazoparib capsules at a dose of 1000 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 1: Talazoparib 1100 mcg/Day: Participants received talazoparib capsules at a dose of 1100 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 2: Talazoparib (Breast Cancer): Participants with breast cancer, received talazoparib capsules at the MTD as determined in Part 1 (1000 mcg/day), orally once daily in each 28-day treatment cycle (up to a maximum of 40 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 2: Talazoparib (Ovarian/ Peritoneal Cancer): Participants with ovarian/ peritoneal cancer, received talazoparib capsules at the MTD as determined in Part 1 (1000 mcg/day), orally once daily in each 28-day treatment cycle (up to a maximum of 40 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 2: Talazoparib (Pancreatic Cancer): Participants with pancreatic cancer, received talazoparib capsules at the MTD as determined in Part 1 (1000 mcg/day), orally once daily in each 28-day treatment cycle (up to a maximum of 40 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 2: Talazoparib (Ewing Cancer): Participants with ewing cancer, received talazoparib capsules at the MTD as determined in Part 1 (1000 mcg/day), orally once daily in each 28-day treatment cycle (up to a maximum of 40 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 2: Talazoparib (SCLC Cancer): Participants with SCLC cancer, received talazoparib capsules at the MTD as determined in Part 1 (1000 mcg/day), orally once daily in each 28-day treatment cycle (up to a maximum of 40 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
- Part 2: Talazoparib (Prostate Cancer): Participants with prostate cancer, received talazoparib capsules at the MTD as determined in Part 1 (1000 mcg/day), orally once daily in each 28-day treatment cycle (up to a maximum of 40 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
Period: Part 1: Dose Escalation
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day | Part 2: Talazoparib (Breast Cancer) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 2: Talazoparib (Pancreatic Cancer) | Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 2: Talazoparib (Prostate Cancer)
Started | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal Cancer | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate Cancer | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ewing Cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic Cancer | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian/ Peritoneal Cancer | 1 | 1 | 2 | 3 | 3 | 4 | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cancer | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 3 | 6 | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 2 | 3 | 2 | 1 | 5 | 5 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Dose Expansion
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day | Part 2: Talazoparib (Breast Cancer) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 2: Talazoparib (Pancreatic Cancer) | Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 2: Talazoparib (Prostate Cancer)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 11 | 12 | 24 | 3
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11 | 10 | 12 | 23 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 10 | 10 | 12 | 24 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 6 | 7 | 11 | 19 | 2
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received at least 1 dose of talazoparib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day | Part 2: Talazoparib (Breast Cancer) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 2: Talazoparib (Pancreatic Cancer) | Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 2: Talazoparib (Prostate Cancer) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 12 | 11 | 10 | 12 | 23 | 3 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (3.51) | 66.7 (9.07) | 64.0 (9.64) | 48.7 (11.50) | 60.7 (5.77) | 61.3 (19.00) | 48.2 (8.66) | 45.0 (18.25) | 38.8 (13.73) | 46.5 (11.47) | 54.2 (10.93) | 65.2 (7.71) | 28.7 (15.18) | 64.0 (10.45) | 57.3 (8.14) | 53.7 (16.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 3 | 3 | 5 | 6 | 5 | 5 | 11 | 11 | 4 | 6 | 11 | 0 | 76
  Male | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 6 | 6 | 12 | 3 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 3 | 6 | 5 | 5 | 4 | 9 | 11 | 10 | 10 | 23 | 3 | 101
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response in participants was defined as the number of participants with complete response (CR) or partial response (PR) after treatment with talazoparib and maintained for at least 4 weeks (28 days) as assessed by response evaluation criteria in solid tumors (RECIST) version 1.1. CR defined as disappearance of all non-nodal target lesions (where all target lesions were recorded with a length of 0 millimeter [mm] on the case report form [CRF]) and the reduction of the shortest diameter of all nodal lesions to less than [<] 10 mm. PR was defined by a 30% or more decrease in the sum of the longest diameters (SLD) + sum of shortest diameters (SSD) of target lesions, taking as reference the baseline SLD+SSD.
Time Frame: From Baseline until disease progression or death due to any cause (maximum duration: 1071 days for Part 1; 834 days for Part 2)
Population: Response analysis population: all enrolled participants who had at least 1 dose of talazoparib, and measurable disease at baseline. Data for this outcome measure was planned to be analyzed combined for Part 1 and Part 2 on the basis of cancer type.
Measure: Number; unit: participants
Groups:
- Part 1 and Part 2: Talazoparib (Breast Cancer): Participants with breast cancer who received talazoparib capsules in Part 1 and 2 at a dose of either 600 mcg/day, 900 mcg/day, 1000 mcg/day, 1100 mcg/day.
- Part 1 and Part 2: Talazoparib (Ovarian/ Peritoneal Cancer): Participants with ovarian/ peritoneal cancer who received talazoparib capsules in Part 1 and 2 at a dose of either 25 mcg/day, 50 mcg/day, 100 mcg/day, 200 mcg/day, 400 mcg/day, 600 mcg/day, 900 mcg/day, 1000 mcg/day, 1100 mcg/day.
- Part 1 and Part 2: Talazoparib (Pancreatic Cancer): Participants with pancreatic cancer who received talazoparib capsules in Part 1 and 2 at a dose of either 25 mcg/day, 50 mcg/day, 1000 mcg/day.
- Part 1 and Part 2: Talazoparib (Ewing Cancer): Participants with ewing cancer who received talazoparib capsules in Part 1 and 2 at a dose of either 1000 mcg/day, 1100 mcg/day.
- Part 2: Talazoparib (SCLC Cancer): Participants with small cell lung cancer (SCLC) cancer who received talazoparib capsules in Part 2 at a dose of 1000 mcg/day.
- Part 1 and Part 2: Talazoparib (Prostate Cancer): Participants with prostate cancer who received talazoparib capsules in Part 1 and 2 at a dose of 600 mcg/day.
- Part 1: Talazoparib (Colorectal Cancer): Participants with colorectal cancer who received talazoparib capsules in Part 1 at a dose of either 25 mcg or 100 mcg/day.
Arm/Group | Part 1 and Part 2: Talazoparib (Breast Cancer) | Part 1 and Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 1 and Part 2: Talazoparib (Pancreatic Cancer) | Part 1 and Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 1 and Part 2: Talazoparib (Prostate Cancer) | Part 1: Talazoparib (Colorectal Cancer)
Number analyzed (Participants) | 20 | 31 | 13 | 14 | 23 | 1 | 2
participants | 8 | 12 | 2 | 0 | 2 | 0 | 0

2. Primary Outcome: Number of Participants With Best Overall Response
Description: Best overall response: best response (in the order of confirmed CR, confirmed PR, stable disease [SD] and progressive disease [PD]) among all overall response as RECIST 1.1, recorded from date of first dose of talazoparib until participant withdrew from study/data cut-off date, whichever earlier. CR defined as disappearance of all non-nodal target lesions (where all target lesions recorded with a length of 0 mm on the CRF) and the reduction of the shortest diameter of all nodal lesions to < 10 mm. PR defined as at least a 30% decrease in sum of the diameters of target lesions, reference to baseline sum diameters. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD defined as at least a 20% increase in sum of diameters of target lesions, reference to the smallest sum on study (this includes the baseline sum if that was the smallest on study).
Time Frame: as for outcome 1
Population: Response analysis population: all enrolled participants who had at least 1 dose of talazoparib, and measurable disease at baseline. Data for this outcome measure was planned to be analyzed combined for Part 1 and Part 2 on the basis of cancer type and was not planned to be analyzed for "Part 1: Colorectal Cancer" arm, as pre-specified in protocol.
Measure: Number; unit: participants
Arm/Group | Part 1 and Part 2: Talazoparib (Breast Cancer) | Part 1 and Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 1 and Part 2: Talazoparib (Pancreatic Cancer) | Part 1 and Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 1 and Part 2: Talazoparib (Prostate Cancer)
Number analyzed (Participants) | 20 | 31 | 13 | 14 | 23 | 1
participants
  Complete Response (CR) | 1 | 1 | 0 | 0 | 0 | 0
  Partial Response (PR) | 7 | 11 | 2 | 0 | 2 | 0
  Stable Disease (SD) | 7 | 10 | 2 | 4 | 4 | 1
  Progressive Disease (PD) | 5 | 6 | 6 | 9 | 14 | 0

3. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time (in weeks) from the date of first dose of study drug to the earlier date of the documented PD or death due to any cause. PD as per RECIST 1.1 defined as at least a 20% increase in the sum of diameters of target lesions, reference to the smallest sum on study (this includes the baseline sum if that was the smallest on study).
Time Frame: Baseline, until PD or death due to any cause (maximum duration:1071 days for Part 1; 834 days for Part 2)
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of talazoparib. Data for this outcome measure was planned to be analyzed combined for Part 1 and Part 2 on the basis of cancer type and was not planned to be analyzed for "Part 1: Colorectal Cancer" arm, as pre-specified in protocol.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1 and Part 2: Talazoparib (Breast Cancer) | Part 1 and Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 1 and Part 2: Talazoparib (Pancreatic Cancer) | Part 1 and Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 1 and Part 2: Talazoparib (Prostate Cancer)
Number analyzed (Participants) | 20 | 34 | 13 | 14 | 23 | 4
weeks | 29.3 [12.1 to 43.4] | 32.1 [18.9 to 38.6] | 5.3 [2.4 to 21.3] | 6.2 [3.1 to 14.0] | 11.1 [4.3 to 13.0] | 12.1 [12.0 to NA]

4. Primary Outcome: Duration of Response
Description: Duration of response was defined as the time (in weeks) from the date of the first documented objective response confirmed at least 28 days later to the date of the first documented PD or date of death, whichever occurred first. PD as per RECIST version 1.1 defined as at least a 20% increase in the sum of diameters of target lesions, reference to the smallest sum on study (this includes the baseline sum if that was the smallest on study).
Time Frame: Baseline until PD or death due to any cause (maximum duration: 1071 days for Part 1; 834 days for Part 2)
Population: Analysis performed on subset of response analysis population which included participants who had objective response. Data for outcome measure was planned to be analyzed combined for Part 1 and Part 2. "Overall number of participants analyzed" is zero (0) for arms of ewing, prostate, CLC cancer, since none of the participants had objective response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part 1 and Part 2: Talazoparib (Breast Cancer) | Part 1 and Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 1 and Part 2: Talazoparib (Pancreatic Cancer) | Part 1 and Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 1 and Part 2: Talazoparib (Prostate Cancer) | Part 1: Talazoparib (Colorectal Cancer)
Number analyzed (Participants) | 8 | 12 | 2 | 0 | 2 | 0 | 0
weeks | 32.2 [20.1 to 64.1] | 26.9 [15.7 to 35.1] | NA [21.6 to NA] — Median and Upper limit of 95% CI were not estimable due to the less number of participants with events |  | 13.6 [12.0 to 15.3] |  |

5. Primary Outcome: Number of Participants With Stable Disease
Description: SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD defined as at least a 20% increase in sum of diameters of target lesions, reference to the smallest sum on study (this includes the baseline sum if that was the smallest on study).
Time Frame: Baseline, until PD or death due to any cause (maximum duration: 1071 days for Part 1; 834 days for Part 2)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Part 1 and Part 2: Talazoparib (Breast Cancer) | Part 1 and Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 1 and Part 2: Talazoparib (Pancreatic Cancer) | Part 1 and Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 1 and Part 2: Talazoparib (Prostate Cancer)
Number analyzed (Participants) | 20 | 31 | 13 | 14 | 23 | 1
participants | 7 | 10 | 2 | 4 | 4 | 1

6. Primary Outcome: Part 1: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose at which no more than 1 of 6 participants experienced a Dose Limiting Toxicity (DLT). DLT defined as any of the following occurring during cycle 1 of part 1 of study, Hematologic toxicity: Any grade 4 or higher hematologic adverse event, Grade 3 thrombocytopenia associated with grade 2 or higher haemorrhage, Grade 3 thrombocytopenia or neutropenia that led to interruption of dosing for 5 or more days. Nonhematologic toxicity: grade 3 or higher laboratory AE which was asymptomatic and rapidly reversible adverse events (returned to baseline or to grade 1 or lower within 7 days), Grade 3 nausea, vomiting, or diarrhea that could be medically managed to grade 2 or lower with anti-emetics and/or anti-diarrheals within 24 hours, Grade 3 fatigue that improved to grade 2 or lower in 5 days or less, Alopecia. Grades based on National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.
Time Frame: Cycle 1 (Day 1 up to Day 42)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of talazoparib.
Measure: Number; unit: mcg/day
Groups:
- Part 1: Talazoparib: All Participants: All participants who received talazoparib capsules in part 1 at a dose of either 25 mcg/day, 50 mcg/day, 100 mcg/day, 200 mcg/day, 400 mcg/day, 600 mcg/day, 900 mcg/day, 1000 mcg/day and 1100 mcg/day once daily from Day 8 to 35 of Cycle 1 and thereafter once daily in each 28-day treatment cycle starting from Cycle 2 (up to a maximum of 50 cycles) until documented disease progression or unacceptable toxicity, or until study discontinuation criteria were met.
Arm/Group | Part 1: Talazoparib: All Participants
Number analyzed (Participants) | 39
mcg/day | 1000

7. Primary Outcome: Part 1: Recommended Part 2 Dose of Talazoparib
Description: The Recommended dose of talazoparib for use in Part 2 was determined in Part 1 (dose escalation) on the basis of the totality of safety, pharmacokinetics (PK), pharmacodynamic and preliminary efficacy data observed in Cycles 1 and 2 and beyond.
Time Frame: Baseline up to Cycle 50 (each cycle 28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of talazoparib.
Measure: Number; unit: mcg/day
Arm/Group | Part 1: Talazoparib: All Participants
Number analyzed (Participants) | 39
mcg/day | 1000

8. Other Pre Specified Outcome: Part 1 and 2: Number of Participants With Treatment-Emergent Adverse Events and Serious Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to end of study (up to 1071 days for Part 1 and up to 834 days for Part 2) that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Part 1: Baseline up to 1071 days; Part 2: Baseline up to 834 days
Population: Safety analyses set included all enrolled participants who received at least 1 dose of talazoparib.
Measure: Number; unit: participants
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day | Part 2: Talazoparib (Breast Cancer) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 2: Talazoparib (Pancreatic Cancer) | Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 2: Talazoparib (Prostate Cancer)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 12 | 11 | 10 | 12 | 23 | 3
participants
  AEs | 2 | 3 | 2 | 3 | 3 | 6 | 6 | 6 | 6 | 12 | 11 | 10 | 12 | 21 | 2
  SAEs | 1 | 2 | 2 | 3 | 0 | 2 | 3 | 1 | 3 | 2 | 5 | 6 | 4 | 8 | 0

9. Other Pre Specified Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Talazoparib
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1 and Day 35
Population: The pharmacokinetic (PK) evaluable population included all participants who received at least 1 dose of talazoparib with adequate PK results to perform PK calculations and was used for analysis of PK endpoints.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
picograms per milliliter (pg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 6
  Cycle 1 Day 1 | 60.0 (15.9) | 79.7 (7.50) | 214 (50.9) | 788 (369) | 1830 (699) | 4100 (1400) | 6100 (3060) | 10600 (4220) | 13200 (3220)
  Cycle 1 Day 35: number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 6 | 5 | 6 | 4
  Cycle 1 Day 35 | 300 (78.8) | 615 (74.2) | 1880 (332) | 5620 (3530) | 6560 (1500) | 11300 (3230) | 15400 (1540) | 21000 (7990) | 23400 (4810)

10. Other Pre Specified Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Talazoparib
Time Frame: Cycle 1 and 2: Predose, 0.5, 1, 2, 3 and 4 hours postdose on Day 1
Population: The PK evaluable population included all participants who received at least 1 dose of talazoparib with adequate PK results to perform PK calculations and was used for analysis of PK endpoints. PK data was planned to be reported for the overall participants in Part 2, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Part 2: Talazoparib 1000 mcg: All participants with either breast, ovarian/peritoneal, pancreatic, ewing, SCLC, or prostate cancer who received talazoparib capsules at a dose of 1000 mcg/day in Part 2.
Arm/Group | Part 2: Talazoparib 1000 mcg
Number analyzed (Participants) | 70
pg/mL
  Cycle 1 Day 1 | 8480 (3890)
  Cycle 2 Day 1: number analyzed (Participants) | 41
  Cycle 2 Day 1 | 17700 (5790)

11. Other Pre Specified Outcome: Part 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Talazoparib
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1 and Day 35
Population: The PK evaluable population included all participants who received at least 1 dose of talazoparib with adequate PK results to perform PK calculations and was used for analysis of PK endpoints.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 6
  Cycle 1 Day 1 | 7.92 [1.95 to 9.95] | 1.00 [0.800 to 1.02] | 1.02 [1.00 to 3.98] | 1.03 [1.00 to 2.32] | 2.03 [0.750 to 2.95] | 0.835 [0.750 to 1.95] | 2.00 [1.02 to 9.98] | 1.03 [0.730 to 2.07] | 1.00 [0.730 to 2.05]
  Cycle 1 Day 35: number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 6 | 5 | 6 | 4
  Cycle 1 Day 35 | 1.02 [0.580 to 3.98] | 5.43 [0.770 to 10.1] | 0.785 [0.750 to 0.820] | 1.97 [1.00 to 3.02] | 0.980 [0.750 to 2.00] | 1.04 [0.730 to 5.98] | 1.02 [0.970 to 2.07] | 1.02 [0.750 to 2.00] | 1.48 [0.980 to 2.00]

12. Other Pre Specified Outcome: Part 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Talazoparib
Time Frame: Cycle 1 and 2: Predose, 0.5, 1, 2, 3 and 4 hours postdose on Day 1
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: Talazoparib 1000 mcg
Number analyzed (Participants) | 70
hours
  Cycle 1 Day 1 | 1.00 [0.500 to 4.07]
  Cycle 2 Day 1: number analyzed (Participants) | 41
  Cycle 2 Day 1 | 1.07 [0.500 to 6.05]

13. Other Pre Specified Outcome: Part 1: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUC0-last) of Talazoparib
Description: Area under the plasma concentration time-curve from zero to the time of last measured concentration (AUC0-last).
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: picograms*hour per mililiter (pg*hr/mL)
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
picograms*hour per mililiter (pg*hr/mL) | 3600 (1360) | 5340 (1960) | 16600 (5320) | 39300 (11700) | 43700 (15000) | 97900 (30000) | 160000 (66100) | 182000 (62400) | 201000 (93400)

14. Other Pre Specified Outcome: Part 2: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUC0-last) of Talazoparib
Description: Area under the plasma concentration time-curve from zero to the time of last measured concentration (AUC0-last).
Time Frame: Cycle 1 and 2: Predose, 0.5, 1, 2, 3 and 4 hours postdose on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Part 2: Talazoparib 1000 mcg
Number analyzed (Participants) | 70
pg*hr/mL
  Cycle 1 Day 1 | 19100 (8850)
  Cycle 2 Day 1: number analyzed (Participants) | 41
  Cycle 2 Day 1 | 50200 (16300)

15. Other Pre Specified Outcome: Part 1: Minimum Observed Plasma Concentration (Cmin) of Talazoparib
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 35
Population: The PK evaluable population included all participants who received at least 1 dose of talazoparib with adequate PK results to perform PK calculations and was used for analysis of PK endpoints. Data for this outcome measure was not planned to be analyzed for Part 2, as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
pg/mL | 169 (58.0) | 299 (133) | 1020 (107) | 2880 (1710) | 2230 (957) | 3470 (1050) | 3180 (802) | 3720 (1590) | 2910 (803)

16. Other Pre Specified Outcome: Part 1: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-inf)] of Talazoparib
Description: AUC (0-inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time.
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
pg*hr/mL | 5330 (1840) | 8320 (1960) | 37600 (6620) | 92700 (48500) | 60100 (15900) | 120000 (26000) | 188000 (85700) | 200000 (64000) | 235000 (111000)

17. Other Pre Specified Outcome: Part 1: Terminal Half-Life (t1/2) of Talazoparib
Description: T1/2 is the time measured for the plasma concentration of talazoparib to decrease by one half.
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1 and Day 35
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 6
  Cycle 1 Day 1 | 100 (11.9) | 129 (42.6) | 229 (158) | 212 (126) | 102 (27.2) | 58.6 (17.3) | 60.4 (10.9) | 52.9 (13.4) | 71.0 (20.6)
  Cycle 1 Day 35: number analyzed (Participants) | 2 | 2 | 2 | 3 | 3 | 6 | 5 | 6 | 4
  Cycle 1 Day 35 | 107 (84.2) | 132 (12.3) | 98.2 (4.83) | 50.9 (19.1) | 90.7 (32.7) | 63.7 (12.7) | 71.0 (14.5) | 50.0 (16.6) | 52.8 (23.2)

18. Other Pre Specified Outcome: Part 1: Apparent Oral Clearance (CL/F) of Talazoparib
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) was influenced by the fraction of the dose absorbed.
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
liter/hour | 5.17 (2.10) | 6.27 (1.66) | 2.72 (0.532) | 2.61 (1.35) | 6.95 (1.71) | 5.19 (0.990) | 5.49 (2.08) | 5.39 (1.59) | 5.32 (1.64)

19. Other Pre Specified Outcome: Part 1: Apparent Volume of Distribution (Vz/F) of Talazoparib
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F was influenced by the fraction absorbed.
Time Frame: Cycle 1: 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 8, 10, 24, 48, 72 and 96 hours postdose on Day 1 and Day 35
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
liter
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 5 | 6
  Cycle 1 Day 1 | 756 (351) | 1240 (742) | 839 (487) | 678 (217) | 1050 (431) | 441 (143) | 468 (169) | 415 (170) | 549 (232)
  Cycle 1 Day 35: number analyzed (Participants) | 2 | 2 | 2 | 3 | 3 | 6 | 5 | 6 | 4
  Cycle 1 Day 35 | 1070 (971) | 1020 (345) | 475 (47.8) | 264 (249) | 818 (326) | 477 (136) | 604 (169) | 373 (144) | 472 (254)

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (maximum duration: 1071 days for Part 1; 834 days for Part 2)
Description: Analysis performed on safety population. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Part 1: Talazoparib 25 mcg/Day | Part 1: Talazoparib 50 mcg/Day | Part 1: Talazoparib 100 mcg/Day | Part 1: Talazoparib 200 mcg/Day | Part 1: Talazoparib 400 mcg/Day | Part 1: Talazoparib 600 mcg/Day | Part 1: Talazoparib 900 mcg/Day | Part 1: Talazoparib 1000 mcg/Day | Part 1: Talazoparib 1100 mcg/Day | Part 2: Talazoparib (Breast Cancer) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) | Part 2: Talazoparib (Pancreatic Cancer) | Part 2: Talazoparib (Ewing Cancer) | Part 2: Talazoparib (SCLC Cancer) | Part 2: Talazoparib (Prostate Cancer)
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/3 | 3/3 | 0/3 | 2/6 | 3/6 | 2/6 | 3/6 | 2/12 | 5/11 | 6/10 | 4/12 | 8/23 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 2/3 | 3/3 | 3/3 | 6/6 | 6/6 | 6/6 | 6/6 | 12/12 | 11/11 | 10/10 | 12/12 | 20/23 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Talazoparib 25 mcg/Day (N=3) | Part 1: Talazoparib 50 mcg/Day (N=3) | Part 1: Talazoparib 100 mcg/Day (N=3) | Part 1: Talazoparib 200 mcg/Day (N=3) | Part 1: Talazoparib 400 mcg/Day (N=3) | Part 1: Talazoparib 600 mcg/Day (N=6) | Part 1: Talazoparib 900 mcg/Day (N=6) | Part 1: Talazoparib 1000 mcg/Day (N=6) | Part 1: Talazoparib 1100 mcg/Day (N=6) | Part 2: Talazoparib (Breast Cancer) (N=12) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) (N=11) | Part 2: Talazoparib (Pancreatic Cancer) (N=10) | Part 2: Talazoparib (Ewing Cancer) (N=12) | Part 2: Talazoparib (SCLC Cancer) (N=23) | Part 2: Talazoparib (Prostate Cancer) (N=3)
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Community acquired infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Talazoparib 25 mcg/Day (N=3) | Part 1: Talazoparib 50 mcg/Day (N=3) | Part 1: Talazoparib 100 mcg/Day (N=3) | Part 1: Talazoparib 200 mcg/Day (N=3) | Part 1: Talazoparib 400 mcg/Day (N=3) | Part 1: Talazoparib 600 mcg/Day (N=6) | Part 1: Talazoparib 900 mcg/Day (N=6) | Part 1: Talazoparib 1000 mcg/Day (N=6) | Part 1: Talazoparib 1100 mcg/Day (N=6) | Part 2: Talazoparib (Breast Cancer) (N=12) | Part 2: Talazoparib (Ovarian/ Peritoneal Cancer) (N=11) | Part 2: Talazoparib (Pancreatic Cancer) (N=10) | Part 2: Talazoparib (Ewing Cancer) (N=12) | Part 2: Talazoparib (SCLC Cancer) (N=23) | Part 2: Talazoparib (Prostate Cancer) (N=3)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 3 | 4 | 3 | 1 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 1 | 1 | 4 | 4 | 2 | 2 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 4 | 4 | 1 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 2 | 4 | 5 | 2 | 1 | 5 | 10 | 4 | 3 | 9 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 2 | 2 | 3 | 3 | 0 | 2 | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 2 | 3 | 3 | 3 | 5 | 1 | 6 | 9 | 4 | 3 | 12 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 2 | 2 | 2 | 1 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 3 | 3 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 3 | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injury corneal (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 1 | 2 | 3 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 3 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 2 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 4 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 3 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 1 | 4 | 5 | 0 | 2 | 4 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 4 | 0 | 0 | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 4 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 3 | 2 | 4 | 0 | 3 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 3 | 1 | 1 | 5 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 3 | 3 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 3 | 0 | 3 | 8 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 5 | 6 | 3 | 5 | 8 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biopsy bone marrow (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Micturition frequency decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adnexa uteri pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Prostatic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 4 | 0 | 5 | 6 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphostasis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast reconstruction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frontal sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.